CLINICAL TRIAL: NCT01092494
Title: Efficacy of Postoperative Cyclic Oral Contraceptive Use After Gonadotropin-releasing Hormone Agonist for the Prevention of Endometrioma Recurrence
Brief Title: Postoperative Cyclic Oral Contraceptive Use for the Prevention of Endometrioma Recurrence
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: DooSeok Choi, Samsung Medical Center
Other Study IDs: 2010-02-020
Record Dates: First submitted 2010-03-23; First posted 2010-03-25 (Estimated); Last update posted 2010-03-25 (Estimated); Status verified 2010-03

CONDITIONS: Endometriosis
Keywords: Endometrioma recurrence; oral contraceptives; gonadotropin-releasing hormone agonist
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- OC use: OC use after postoperative gonadotropin-releasing hormone agonist treatment
- OC non-use: Only postoperative gonadotropin-releasing hormone agonist treatment

SUMMARY:
Ovarian endometriotic cyst (endometrioma) is one of the most common endometriotic lesions, and conservative laparoscopic surgery is the treatment of choice. However, the recurrence after surgery is common.

As repetitive surgery leads to morbidities and ovarian function decrease, recurrence after surgery frustrates both patients and clinicians. In this aspect, medical treatments have been offered after surgery to prevent or delay the recurrence. Gonadotropin-releasing hormone agonist (GnRHa) is frequently used in women with advanced endometriosis, but the efficacy is rather controversial. On the other hand, it has been demonstrated that oral contraceptives (OCs) could reduce or delay endometrioma recurrence, but data are still limited. Consequently, no one type of postoperative medical therapy has been shown to be superior in reducing the recurrence of endometrioma.

The rationale of postoperative medical therapy is that it could eradicate microscopic lesions which were not found and not treated sufficiently during surgery. Therefore, the maintenance of strongly suppressed condition induced by postoperative GnRHa treatment by addition of OCs could be a promising treatment to prevent the recurrence, but it has not been widely investigated.

We performed this retrospective cohort study to evaluate the efficacy of cyclic monophasic low-dose OCs as a maintenance therapy after GnRHa treatment for the suppression of endometrioma recurrence.

ELIGIBILITY:
Inclusion Criteria:

1. reproductive aged women who underwent conservative laparoscopic ovarian surgery for endometrioma (ASRM stage III/IV) which was confirmed by pathologic inspection
2. women who were given postoperative GnRHa injections every 28 days for 3 or 6 months
3. women with no residual lesion confirmed by ultrasonography after surgery
4. women who were followed up for over 12 months after surgery.

Exclusion Criteria:if they had

1. undergone hysterectomy during an operation
2. been given GnRHa injections more than 6 times
3. been given other types of postoperative treatment (progestin or intrauterine device)
4. a history of previous pelvic surgery for endometriosis
5. a history of hormonal treatment before surgery
6. been diagnosed as menopause after surgery
7. contraindications to OCs
8. been identified ovarian endometriomas within 6 months of postoperative evaluation

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Reproductive aged women who underwent conservative laparoscopic surgery for ovarian endometrioma and followed up at Samsung Medical Center between January 2000 and December 2007.
Sampling Method: Non-Probability Sample
Enrollment: 232 (Estimated)
Dates: Start 2010-03; Primary Completion 2010-03 (Estimated); Study Completion 2010-03 (Estimated)

PRIMARY OUTCOMES:
recurrence rate of endometrioma | 60 months

CONTACTS AND LOCATIONS:
Overall Officials: DooSeok Choi, Study Director — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, Seoul, South Korea

REFERENCES:
- [Background] Park HJ, Koo YA, Yoon BK, Choi D. Postoperative long-term maintenance therapy with oral contraceptives after gonadotropin-releasing hormone analog treatment in women with ovarian endometrioma. J Minim Invasive Gynecol. 2009 Jan-Feb;16(1):34-9. doi: 10.1016/j.jmig.2008.09.582. Epub 2008 Oct 30. PMID 18976968